CLINICAL TRIAL: NCT07375342
Title: Effect of Preoperative Oral Melatonin on Emergence Agitation Following Pediatric Tonsillectomy: a Randomized Controlled Trial
Brief Title: Melatonin for Post Tonsillectomy Emergence Agitation in Pediatric
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Taghreed Elshahat Sakr, lecturer of anesthesia and icu, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RC.2.11.2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Post Tonsillectomy Emergence Agitation
Keywords: agitation; tonsillectomy; pediatric
MeSH Terms: conditions — Psychomotor Agitation | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Melatonin Group) (Active Comparator)
  Interventions: Drug: Melatonin
- Group P (Placebo Group) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Participants will receive Oral melatonin at a dose of 0.5 mg/kg (maximum 20 mg) administered 30 minutes before induction of anesthesia. Dose chosen based on prior pediatric studies and safety data. The tablet will be crushed and mixed with a small amount of water or juice to facilitate administration,
  Arms: Group M (Melatonin Group)
Drug: Placebo — Participants will receive an identical placebo tablet administered 30 minutes before induction of anesthesia.
  The tablet will be crushed and mixed with a small amount of water or juice to facilitate administration,
  Arms: Group P (Placebo Group)

SUMMARY:
The goal of this clinical trial is to learn if melatonin can decrease emergence agitation in pediatric post tonsillectomy. The main questions it aims to answer are:

Does melatonin decrease emergence agitation in pediatric post tonsillectomy? What medical problems do participants have when taking melatonin? Researchers will compare melatonin to a placebo (a look-alike substance that contains no drug) to see if melatonin works todecrease emergence agitation in pediatric post tonsillectomy

Participants will receive Oral melatonin at a dose of 0.5 mg/kg (maximum 20 mg) administered 30 minutes before induction of anesthesia. Dose chosen based on prior pediatric studies and safety data.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II.
* Parent/legal guardian provides written informed consent

Exclusion Criteria:

* • Known allergy or contraindication to melatonin.

  * Pre-existing neurological or psychiatric disorders (e.g., epilepsy, autism, ADHD).
  * Children receiving any sedative or psychoactive medication within 48 hours of surgery.
  * Emergency surgery or any procedure other than tonsillectomy/adenoidectomy.
  * Children with known sleep disorders or those taking melatonin supplements.
  * Developmental delay, neurologic disorders, sleep disorders, or known obstructive sleep apnea requiring ICU postoperatively.
  * Hepatic or renal dysfunction (ALT/AST >2×ULN, Cr >1.5 mg/dL)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Emergence Agitation (EA): EA will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale | 5, 10, 15, and 30 minutes after arrival in the PACU.
  The PAED scale consists of five items (eye contact, awareness of surroundings, purposeful actions, restlessness, and inconsolability), each scored from 0 to 4. Total score ranges from 0 to 20., scale ≥10 or equivalent define the presence of clinically significant EA

SECONDARY OUTCOMES:
Time to Discharge | 10-30 min from arriving to PACU
  Measured as the time from PACU arrival to achieving a modified Aldrete score (a 10-point system used in the post-anesthesia care unit (PACU) to assess a patient's recovery and determine if they are ready for discharge. It evaluates five categories: Activity, Respiration, Circulation, Consciousness, and Oxygen saturation. Each category is scored from 0 to 2, and a total score of 9 or 10 generally indicates that the patient can be safely discharged from the PACU). ≥9 (min),
Postoperative Pain | first 2 hours postoperative
  Assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) scale at the same time points as the PAED scale.
Rescue Analgesia | 24 hours after surgery
  Total dose of rescue analgesia (e.g., intravenous morphine or fentanyl measured according to the child weight in kg ) required in the PACU.
Adverse Events | first 24-hour post operative
  Incidence of PONV, respiratory depression (defined as {SpO}_2 < 90% requiring intervention), bradycardia (<60 bpm), intraoperative hemodynamic instability excessive sedation (Ramsay Sedation Scale > 3) and other adverse events.
Parent/caregiver satisfaction | first 24-hour post operative
  measured at discharge (Likert scale) used to measure attitudes, opinions, and behaviors by asking respondents to rate their level of agreement or intensity of feeling regarding a statement, it include options such as strongly disagree, disagree, somewhat disagree, either agree or disagree, somewhat agree, and agree

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No